CLINICAL TRIAL: NCT05423301
Title: Impact of Global Physiotherapy on Acute Respiratory Failure Within 7 Days After Extubation in Intensive Care Unit Patients With High Risk of Extubation Failure.
Brief Title: Global Physiotherapy in ICU Patients With High Risk Extubation Failure
Acronym: KINEXTUB
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CHUBX 2020/51
Record Dates: First submitted 2022-06-14; First posted 2022-06-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Acute Respiratory Failure
Keywords: Physiotherapy; Intensive care unit; Extubation; High-risk patients; Acute respiratory failure

STUDY DESIGN:
Intervention Model Description: The proposed study will be a single-center open-label comparative randomized clinical study, in two parallel arms, at the Bordeaux University Hospital. Patients extubated during working hours on Mondays to Friday in the presence of the physiotherapy team will be included in the study and randomized with a 1: 1 ratio between the experimental arm and the control arm. In both groups, patients are routinely alternated between high-flow oxygenation and NIV, adjusted to patient-specific goals, as recommended for these patients.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental (Experimental)
  Interventions: Procedure: Experimental
- control (Active Comparator)
  Interventions: Procedure: Control

INTERVENTIONS:
Procedure: Experimental — Respiratory care consists of manual and instrumental bronchial clearance techniques: Expiratory Flow Enhancement (EFE), suctioning, manual cough assist techniques, instrumental clearance techniques (suctioning and Cough Assist) and swallowing disorder management.)
  Arms: experimental
Procedure: Control — The control group will receive early respiratory care and rehabilitation by nurses, nurses' aides and doctors until D7. Respiratory care includes aerosol therapy, oral and pharyngeal clearance with aspirations, verbal coughing and sputum removal, and possibly bronchial fibroscopy for clearance if necessary. Early rehabilitation consists of alternating postures in bed, passive chair positioning (patient lift), or active positioning via a bed rail and standing.
  Arms: control

SUMMARY:
This study aims to compare care provided by physiotherapists, combining respiratory care and early rehabilitation in intensive care unit, with standard care on the rate of acute respiratory failure within 7 days after extubation, in patients with high risk of extubation failure.

DETAILED DESCRIPTION:
The extubation failure rate is 15% on average in intensive care units, but can reach 30% within 48 hours after extubation in high risk patients. Their characteristics are : age > 65 years, respiratory disease, body mass index > 30 kg / m², intubation for more than 7 days, first extubation failure, and patient with ineffective cough associated with bronchial obstruction. The main reason for reintubation in these patients is acute respiratory failure with an ineffective cough, a bronchial obstruction, and neuromyopathy. On these three components, the physiotherapist can apply specific techniques. Even though scientific literature recommends the presence of a physiotherapist before, during and after extubation in patients intubated for more than 48 hours, the benefits of physiotherapy in this context remains poorly explored.

The main objective of this study is to compare the rate of acute respiratory failure within 7 days post-extubation in high-risk intensive care patients. The secondary objectives are to compare the ROX index, the reintubation rate for acute respiratory failure within 7 days after extubation, the rate of pneumonia at 7 days, time spent on respiratory and mobilization care.

ELIGIBILITY:
Inclusion Criteria:

* Patients with spontaneous ventilation weaning test.
* Consent form signed by the person support.

Exclusion Criteria:

* Patients with a self-extubation,
* Patients with a tracheostomy,
* Patients with acute respiratory failure for acute lung edema (OAP),
* Patients with decision to limit or stop Active Therapeutics (LATA).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Estimated)
Dates: Start 2023-10-03 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Rate of acute respiratory failure | During 7 days post extubation
  The primary endpoint is the proportion of patients with post-extubation acute respiratory failure, defined as the occurrence within 7 days of extubation of at least two of the following criteria: respiratory acidosis (pH <7.35, PaCO2 >45 mmHg), hypoxemia (PaO2 <60 mmHg with a FiO2 >40% or PaO2/FiO2<150) and respiratory rate >35/min.

SECONDARY OUTCOMES:
ROX index | 8 hours during 7 days post extubation
  ROX index is calculated every 8 hours during the 7 days post-extubation, ROX index is defined by the ratio of oxygen saturation measured by pulse oximetry/FiO2 to respiratory rate.
Rate of reintubation | During 7 days post extubation
  The rate of reintubation within 7 days post-extubation, with reintubation occurring contemporaneously with the onset of acute respiratory failure, without expected clinical improvement,
Rate of pneumopathy | During 7 days post extubation
  Lung disease is defined by the following criteria:
  o Radiological signs : Two successive films from which the appearance of a focus of lung disease is suspected, If there is no history of heart or lung disease: one scan is sufficient.
  o At least one of the following signs: temperature > 38.5° without other cause leukocytes < 4000/mm3 or > 12000/mm3
  o And at least two of the following signs: Purulent secretions Cough or dyspnoea Desaturation or increased oxygen requirement or need for ventilatory support
Time for respiratory care | During 7 days post extubation
  The mean time spent on respiratory care or mobilisation of patients estimated daily in the 7 days following extubation. Time estimated in minutes.

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux - Hopital Haut-Lévêque, Pessac, France